CLINICAL TRIAL: NCT01598636
Title: The Lateral Tibial Tunnel in Anterior Cruciate Ligament Surgery. A Clinical and Ct-graphic Study.to Evaluate the Concept
Brief Title: The Lateral Tibial Tunnel in ACL Surgery
Acronym: LTT-HVDB
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); GZA Ziekenhuizen Campus Sint-Augustinus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012/324
Record Dates: First submitted 2012-05-09; First posted 2012-05-15 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Anterior Cruciate Ligament Revision Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lateral Tibial Tunnel technique (Experimental)
  Interventions: Procedure: Lateral tibial tunnel

INTERVENTIONS:
Procedure: Lateral tibial tunnel — To reduce the rehabilitation time after ACL revision surgery due to a better surgical technique

SUMMARY:
The Lateral Tibial Tunnel technique is a new concept in Anterior Cruciate Ligament (ACL) surgery. In this technique a tibial tunnel is drilled from the antero-lateral side of the tibia towards the ACL footprint. This technique allows the surgeon to deal with bone stock problems in the antero-medial part of the tibia as often encountered in ACL revision surgery. In ACL revision surgery it is often impossible to perform a one-stage revision surgery procedure due to bone stock deficiency in the antero-medial side of the tibia. It is hypothesized that the Lateral tibial tunnel technique allows the surgeon to perform a one-stage procedure instead of a two stage procedure. Furthermore the lateral tibial tunnel technique allows better graft fixation in two-stage ACL revision surgery. Several biomechanical studies proved biomechanical superiority of the new technique compared to the classical technique.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring ACL revision surgery
* patients requiring ACL surgery who have bone stock problems at the medial side of the proximal tibia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of clinical scores pre-operative | pre-operative
evaluation of clinical scores at 3 months | 3 months post operative
Evaluation of clinical scores at 6 months | 6 months post operative
Evaluations of clinical scores at 1 year | 1 year post operative
Evaluation of CT scan and X-ray pre-operative | pre-operative
Evaluation of CT scan and X-ray post-operative | post-operative
Evaluation of CT scan and X-ray 1 year post-operative | 1 year post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Peter Verdonk, MD, Phd, Principal Investigator — University Hospital, Ghent
Locations (3):
- Belgium (3):
  - GZA Sint-Augustinus, Antwerp
  - University Hospital, Ghent
  - University Hospital, Leuven

REFERENCES:
- See also: Related Info — http://www.uzgent.be